CLINICAL TRIAL: NCT06962358
Title: Three Years Radiographic Evaluation of Different Implant Retained Complete Over Denture Attachments (In Vivo Study)
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nashwa ali saleh, Principlae investigator, Tanta University
Other Study IDs: (#R-RP-2-24-3163).
Record Dates: First submitted 2025-04-23; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Treatment of Fully Edentoulous Patients
Keywords: Implant; Over denture; Attachment; Preapical radiograph

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abstract: Treatment of completely edentulous patients with implant over dentures became a common treatment modality that greatly improves the patient's quality of life. AIM: The aim of this randomized clinical trial was to evaluate three different types of implants retained over denture attachment for three years of fellow up. Material and Methods: In a randomized prospective trial 24 completely edentulous patients of age ranged from 50-65 years were carefully selected. The patients were divided into 3 groups group A patients of implant retained over denture with telescopic attachment, Group B patients of implant retained over denture with locator attachment and Group C implant retained over denture with ball and socket attachment, over three years radiographic evaluation was carried out

DETAILED DESCRIPTION:
According to Zarb el al., 15acrylic denture was constructed first Then a radiographic template was prepared16. Two separate CBCT (dual scan technique) images of the radiographic stent were acquired using a CAT FLX V17, Nc 28273, Kavo, Charlotte, USA. data acquired from DICOM Superimposition in implant planning software (In2guide by 3DIEMME) ® allowed for precise evaluation of implant sites in edentulous regions (virtual placement of implants considering the relation to anatomical structures and prosthetic requirements) since the prosthesis could be seen over the accessible bone architecture. , Two implants positioned vertically (Narrow sky 3512, bredent, Germany) for all patients Two healing abutments were screwed into place after the canine regions were bilaterally implanted with narrow plate forms measuring 3.5 mm in diameter and 12 mm in length. The denture was put back into place with silicon soft lining materials after 7 days of healing, and it was meant to be worn for one month. Patients who got telescopic attachments for their implant-retained overdentures were randomly assigned to one of three groups of eight patients each based on GA. (GB): the individual who got an implant-retained overdenture that has a locator attachment (Gc): the individual who got an implant-retained overdenture that has a ball and socket fixation

ELIGIBILITY:
Inclusion CritThe inclusion criteria of the study:

1. Patients who have no teeth have been at least six months since their last extraction
2. Having no underlying health conditions that could slow or prevent the repair of soft or hard tissues
3. Cone-beam computed tomography (CBCT) confirms that each patient has an adequate amount and quality of remaining alveolar bone,
4. Patients should have generally good dental hygiene
5. They should have an Angel class I maxillomandibular relation with at least 20 mm of inter-arch space for telescopic attachment, and 6. mm of residual alveolar bone width in the mandibular canine sections.

eria:

-

Exclusion Criteria:

* The exclusion criteria of the study:

  1. A patient who has already undergone radiation treatment to the neck and head area.
  2. With the present steroid treatment
  3. If they have a mental or neurological disability that could make it difficult for them to practice proper dentist care.
  4. When a person's immune system is weak.
  5. I have developed parafunctional behaviors.
  6. In cases where the patient is highly sedentary, frequently smokes, or otherwise refuses to cooperate with treatment.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Using a permuted block randomization procedure, patients were selected at random. By utilizing sealed envelopes, the individual responsible for assigning participants to the intervention arm remained oblivious to the allocation sequence and code. Somebody other than the people who took part in the study made this choice.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation | 3 year
  (a) In periapical radiographs, by using Digora software (DIGORA. ® for Windows2.7. SOREDEX, Finland.) the distance from the marginal osseous level to the implant platform was measured in millimeters,22 in mesial and distal aspects of each implant. During the implant platform selection process, two reference sites were made that could be readily seen and located. At a height of zero, we used a straight line that connected the two spots as our reference. Starting at zero height and continuing distally to the implant, a perpendicular line was drawn to determine the bone level. The line was then used to measure the distance from the implant to the bone.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta unversity, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided